CLINICAL TRIAL: NCT06972953
Title: NEUROvascular NAVigation With Remotely Controlled Deflectable Guidewire, Study I (NeuroNAV Study I)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artiria Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FR 2024
Record Dates: First submitted 2025-05-02; First posted 2025-05-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Unruptured Cerebral Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SmartGUIDE (deflectable guidewire) (Experimental)
  Interventions: Device: SmartGUIDE (deflectable guidewire)
- Any standard of care guidewire (Active Comparator)
  Interventions: Device: Any standard of care guidewire

INTERVENTIONS:
Device: SmartGUIDE (deflectable guidewire) — SmartGUIDE is a deflectable guidewire for use in interventional procedures in the neurovasculature and the peripheral vasculature. It can be used to selectively introduce and position catheters and other interventional devices within the peripheral and neurovasculature. The device is a steerable guidewire with a deflectable tip. This allows adjusting the shape of the tip, dynamically, while the physician navigates the device in the patient's arterial and venous circulatory system.
  Arms: SmartGUIDE (deflectable guidewire)
Device: Any standard of care guidewire — The control device is any standard of care guidewire as per hospital routine indicated for neuro-interventional procedures.
  Arms: Any standard of care guidewire

SUMMARY:
The aim of the study is to confirm the safe and successful use of the SmartGUIDE guidewire, when used in neuro interventions. The performance of the SmartGUIDE guidewire in terms of safe and successful navigation within the neurovasculature will be compared to standard of care guidewire on the market.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Informed consent signed by the patient
* Confirmed cerebral unruptured aneurysm treatable via transcatheter approach

Exclusion Criteria:

* Pregnancy or lactation
* Known disorder of vascular fragility with propensity to vascular injury (e.g., Ehlers-Danlos syndrome)
* Known prior vascular stenosis or dissection or injury to vessels intended to be catheterized during study procedures
* Acute phase myocardial infarction or uncontrolled cardiac arrhythmia
* Uncontrolled serum electrolyte imbalance
* Bleeding disorder which limits the use of antiplatelet and/or anticoagulant therapy
* Known contraindication to intravascular contrast material that cannot be adequately controlled with pre-medication
* Known hypersensitivity to Nickel
* Subjects currently enrolled in another investigational device or drug study that clinically interferes with the current study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Performance | During index procedure
  Intra-procedural technical success defined as successful navigation of device to the target vessel without need for shaping by hand, removal or exchange.

SECONDARY OUTCOMES:
Usability | During index procedure
  Usability data (shape retention, pushability, trackability, navigability, support, proximal access complexity) collected through questionnaire.
Procedural times | During index procedure
  Procedural times (duration of tip reshaping, duration of access to target, duration of fluoroscopic exposition).
Intra-procedural adverse events | During index procedure and up to 48 hours post procedure
  Occurrence of adverse events.
Intra-procedural device deficiencies | During index procedure
  Occurrence of intra-procedural device deficiencies.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Aymeric Rouchaud, Principal Investigator — Centre Hospitalier Universitaire - CHU Limoges
Locations (1):
- Centre Hospitalier Universitaire - CHU Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No